CLINICAL TRIAL: NCT06155253
Title: Comparing Analgesic Efficacy and Quality of Recovery of Bi-level and Single-level Erector Spinae Plane Block for Open Inguinal Hernia Repair Surgery - a Randomised, Observed-blinded Active-controlled Trial
Brief Title: Comparing Bi-level and Single-level ESP Block for Open Inguinal Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Patricia Ip, Resident, Hospital Authority, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIRB-2023-091-2
Record Dates: First submitted 2023-10-19; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Hernia, Inguinal
Keywords: open inguinal hernia repair; erector spinae plane block; multi-level; bi-level; single-level; single-injection
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-level ESP group (1ESP) (Active Comparator): Subjects in 1ESP group will receive a single-shot single-level erector spinae plane block at L1 level under ultrasound guidance immediately before surgery.
  Interventions: Procedure: Erector spinae plane block
- Bi-level ESP group (2ESP) (Active Comparator): Subjects in this group will receive a single-shot single-level erector spinae plane block at T12 and L1 levels under ultrasound guidance immediately before surgery.
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — ESP block is a paraspinal fascial plane block that involves injection of local anesthetic underneath the anterior fascia of the erector spinae muscles.
  Local anaesthetic mixture (lignocaine 2% with adrenaline, bupivacaine 0.25%) will be delivered with insulated needle in bolus(es) to above-mentioned levels (L1 in 1ESP group, T12 & L1 in 2ESP group)

SUMMARY:
The goal of this clinical trial is to compare the effects of single-level and bi-level erector spinae plane block in open inguinal hernia repair surgery. The main question it aims to answer are:

* Whether bi-level ESP block will improve pain control after open inguinal hernia repair surgery
* Whether bi-level ESP block will improve quality of recovery after open inguinal hernia repair surgery

Participants will receive erector spinae plane block, and will be randomised into 2 groups, single-level ESP block and bi-level ESP block, before open hernia repair surgery. They will be followed up after operation for assessment of pain control and quality of recovery.

DETAILED DESCRIPTION:
Open inguinal hernia repair is increasingly performed as a day case surgery. As a result, satisfactory acute pain control is very important to reduce discomfort, as well as to facilitate early mobilisation and recovery. Regional anaesthesia, eg. erector spinae plane block (injection below para-spinal muscles) is increasingly implemented as part of multi-modal analgesia to establish better post-operative pain control and spare the use of opioids which can lead to unwanted side effects eg. sedation, nausea and vomiting. Acute post-surgical pain from open inguinal hernia repair consists of subcutaneous, deep somatic and visceral components. The erector spinae plane (ESP) block acts by local anaesthetic (LA) spread to ventral and dorsal rami of spinal nerves, producing somatic and visceral pain relief. Therefore, it can effectively relieve acute post-surgical pain resulted from open hernia repair. Bi-level ESP block has been utilised clinically to provide multi-dermatomal analgesia in pain management eg. flail chest; or anaesthetic management eg. open inguinal hernia repair, scoliosis surgery, mastectomy. However, to date, there have been no studies comparing the analgesic efficacy of bi-level and single-level erector spinae plane blocks. The investigators postulate that comparing with single-level ESP block, bi-level ESP block can facilitate LA spread into paraspinal areas more effectively, producing more reliable analgesia; and therefore would reduce post-operative pain scores and improve quality of recovery in patients undergoing open inguinal hernia repair.

To investigate the above clinical question, a parallel-group observer-blinded randomised clinical trial was designed. Patients will be randomised into 2 groups. One group of patients (2ESP) will receive ESP block at ipsilateral T12 and L1; while the other group of patients (1ESP) will receive ESP block at ipsilateral L1. L1 was chosen as an injection level, since it is at the midpoint of corresponding spinal nerve roots innervating the groin (T12-L3). For bi-level injection group, thoracic instead of another lower lumbar level was chosen to avoid motor blockade caused by excessive local anaesthetic spread into lumbar plexus, leading to delayed mobilisation which is undesirable for patients undergoing ambulatory surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years old
* ASA (American Society of Anesthesiologists) class I to III
* Unilateral open inguinal hernia repair

Exclusion Criteria:

* Patient refusal or unable to consent to study
* Contraindication of ESP block including patient refusal, injection site infection, coagulopathy, hypersensitivity to local anaesthetic
* Pre-existing chronic pain
* Alcohol and substance dependence
* Pre-existing psychiatric diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain score | 1 day
  Numeric rating score (11-point scale) will be used to assess pain. (0 = no pain, 10 = worst pain)
Quality of recovery score (QoR-15) | 1 day
  This is a validated questionnaire to evaluate the physical, emotional and functional aspects of patients and their abilities to resume usual activities of daily living after surgery and anaesthesia. It ranges from 0-150. Higher score indicates better recovery.

SECONDARY OUTCOMES:
Peri-operative fentanyl dosage | 1 day
  Dosage of fentanyl in micrograms used in the peri-operative period will be compared between both groups.
Time to first rescue analgesic | 1 day
  Time from completion of ESP block to first rescue analgesic will be recorded and compared.
Rate of motor deficit | 1 day
  Rate of lower limb weakness in both groups of subjects affecting ambulation / weight bearing will be compared.
Rate of post-operative urinary retention | 2 days
  Rate of post-operative urinary retention in both groups of subjects affecting gait / weight bearing will be compared.
Rate of post-operative nausea and vomiting | 2 days
  Rate of post-operative nausea and vomiting in both groups of subjects will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Ip, Principal Investigator — HA